CLINICAL TRIAL: NCT06010212
Title: Fruquintinib Combined With Camrelizumab, Paclitaxel Liposome and Nedaplatin as First Line Treatment in Patients With Recurrent Esophageal Squamous Cell Carcinoma
Brief Title: Fruquintinib as First Line Treatment in Patients With Recurrent Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-013-CH11 IIT-ESCC
Record Dates: First submitted 2023-08-09; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Fruquintinib ，Carrelizumab，Advanced ESCC
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; nedaplatin; HMPL-013

STUDY DESIGN:
Intervention Model Description: Fruquintinib,Camrelizumab, Paclitaxel liposome combined with nedaplatin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Fruquintinib,Camrelizumab, Paclitaxel liposome combined with nedaplatin
  Interventions: Drug: Fruquintinib Combined With Camrelizumab, Paclitaxel Liposome and Nedaplatin

INTERVENTIONS:
Drug: Fruquintinib Combined With Camrelizumab, Paclitaxel Liposome and Nedaplatin — Phase Ib: Patients with advanced ESCC will be enrolled in a 3+3 dose escalation fashion, with projected enrolment of between 9-18 patients to determine RP2D. Once the RP2D is confirmed, the study will proceed to phase II.
  fruquintinib: 3 mg, 4 mg, or 5 mg qd p.o., 2 weeks and 1 week, every 3 weeks ( dose exploration phases were performed sequentially from the 4 mg group, refer to the study design section for specific protocols); Camrelizumab: 200 mg I.V D1, every 3 weeks for treatment cycles; Paclitaxel liposomes: 135 mg/m2 i.v d1, administered every 3 weeks, up to 6 cycles; Nidaplatin: 70 mg/m2 i.v d1, administered every 3 weeks, up to 6 cycles. Chemotherapy is used for up to 6 cycles, followed by maintenance therapy with fruquintinib + Camrelizumab until disease progression or intolerable toxicity.
  Phase II: Up to a total of 30 patients with advanced ESCC will be enrolled.
  Other Names: Fruquintinib, Camrelizumab, Paclitaxel liposome combined with nedaplatin

SUMMARY:
This Study is a Single-center, Single-arm, Phase II Clinical Study. The Primary Objective is to Evaluate the Efficacy and Safety of Fruquintinib, Carrelizumab, Paclitaxel Liposomes combined with Nidaplatin as First-line Treatment in Advanced Esophageal squamous cell carcinoma .

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily to join the study and sign the informed consent form;
2. Male or female patients aged 18-70 years (inclusive);
3. Histological or cytology-confirmed unresectable advanced or metastatic ESCC;
4. Identify at least one measurable lesion that meets the requirements of Efficacy Evaluation Criteria for Solid Tumors (RECIST) version 1.1; If a lesion that has previously received local therapy (radiotherapy, ablation, vascular intervention, etc.) is the only lesion, there must be a clear radiographic basis for disease progression of that lesion;
5. Previous systemic therapy for advanced ESCC;
6. ECOG ≤2;
7. Laboratory tests: neutrophil ≥ 1.5×109/L; platelets≥ 75×109/L; Hemoglobin≥ 90g/L; Serum creatinine ≤ 1.5 times the upper limit of normal and creatinine clearance ≥ 60 ml/min; Urine protein <2+; If the urine protein ≥ 2+, the 24-hour urine protein should be < 1 g; Alanine aminotransferase and glutamate aminotransferase ≤ 1.5 times the upper limit of normal, or 3 times the upper limit of normal in the presence of liver metastases≤; total bilirubin ≤ 1.5 times the upper limit of normal or 3 times the upper limit of normal in the presence of liver metastases≤; albumin≥ 3.0 g/dL; Coagulation function: prothrombin time (PT), international normalized ratio (INR) ≤ 1.5x ULN;
8. Female patients with negative urine or blood hCG (except menopause and hysterectomy), female patients of childbearing age and their partners take effective contraceptive measures during the trial and within 3 months after the end of the last dose (e.g., combination of hormones (including estrogen and progesterone) combined with ovulation suppression, progestogen contraception combined with ovulation suppression, intrauterine device, intrauterine hormone release system, bilateral tubal ligation, vasectomy, avoidance of sexual behavior, etc.)

Exclusion Criteria:

1. Known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components, or known to be allergic to fruquintinib or paclitaxel liposomes or nidaplatin components;
2. Have a second tumor within the past 5 years, except cured basal cell carcinoma of the skin or squamous cell carcinoma of the skin or carcinoma in situ of any other site;
3. Uncontrolled serious medical diseases that the investigator believes will affect the patient's ability to receive treatment with the study protocol, such as serious medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled infection, etc.;
4. The patient currently has gastrointestinal diseases such as active gastric and duodenal ulcer and ulcerative colitis, or active bleeding in unremoved tumors, or other conditions that may cause gastrointestinal bleeding and perforation as determined by the investigator; or those who have previously had gastrointestinal perforation or gastrointestinal fistula, which has not recovered after surgical treatment;
5. Patients with evidence of bleeding tendency or history (such as melena, hematemesis, hemoptysis, bloody stools, etc.) within 2 months before the first dose;
6. During screening, it was found that the tumor invaded the structure of large vessels, such as pulmonary artery, superior vena cava or inferior vena cava, etc., and the investigator judged that there was a greater risk of bleeding;
7. History of arterial thrombosis or deep vein thrombosis within 6 months before the first dose; or a stroke event and/or transient ischaemic attack within 12 months; Thrombosis due to implantable intravenous infusion pump or catheter-derived thrombosis, or superficial vein thrombosis, except for those with stable thrombosis after conventional anticoagulation therapy;
8. Receiving chemotherapy, targeting, immunotherapy, clinical trials, etc. of other investigational drugs within 4 weeks before the administration of the first treatment;
9. Patients previously diagnosed with coronary heart disease or ischemic cerebrovascular disease;
10. Pregnant or lactating female patients;
11. Have any other disease, metabolic disorder, abnormal result of physical examination or laboratory test and have reason to suspect that may contraindicate the use of the test drug, or affect the reliability of the results of the study;
12. Undergone major surgery within 28 days before the first dose, or received radiotherapy within 14 days before the first dose, or used radiation agents (strontium, samarium, etc.) within 56 days before the first dose;
13. Judged by the investigator to be unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR（Objective response rate） | 1 year
  Objective Response Rate (ORR) is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions.

SECONDARY OUTCOMES:
DCR（Disease control rates） | 1 year
  Disease Control Rate (DCR) is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) or stable disease (SD) based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
PFS（Progression-free survival） | 1 year
  PFS is defined as the proportion of patients without disease progression (PD or relapse from CR) or death due to any cause at 6 months. Disease progression will be assessed using RECIST (version 1.1). Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Gu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
Plan to publish papers in 2025.